CLINICAL TRIAL: NCT00947258
Title: Influence of Stretching Hamstring and Quadriceps Femoral Muscles on Peak Torque and the Maximum Power of the Knee
Brief Title: Influence of Stretching on Muscle Performance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fortaleza University (Other)
Allocation: Randomized | Masking: Single | Purpose: Prevention
Other Study IDs: 01
Record Dates: First submitted 2009-07-27; First posted 2009-07-28 (Estimated); Last update posted 2009-07-28 (Estimated); Status verified 2009-07

CONDITIONS: Muscle Strength
Keywords: Muscle Strength; Torque; Muscle Stretching Exercises; Range of Motion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Stretching — Participants were divided into 3 groups. The group was referred to stretching 3 weekly for 4 consecutive weeks. Group B went 4 weeks without any intervention and held only one stretch before the re-test. And the group C performed passive knee mobilization. All participants were assessed for goniometry of the knee in flexion and extension and peak torque and power on the isokinetic dynamometer.
  Other Names: peak of torque; performance; isokinetic dynamometer

SUMMARY:
The stretching is performed within sports to improve muscle performance and prevent muscle injury. However, recent studies are contradictory with common practice. Then raised the possibility that stretching before physical activity performed can decrease the muscle performance of healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 30 years.
* History of at least 3 months without performing any physical activity

Exclusion Criteria:

* Recent history of injuries in lower limbs.
* Contraindication to agree with the Par-Q form.
* Make physical activity during the search
* Fails every session of stretching
* BMI above 28
* Pain in the lumbar spine
* I had muscle shortening in Test Thomas (TT) and / or test the popliteal angle (TAP)

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15

CONTACTS AND LOCATIONS:
Locations (1):
- Gabriel Peixoto Leão Almeida, Fortaleza, Ceará, Brazil

REFERENCES:
- See also: Related Info — http://www.unifor.br/coetica